CLINICAL TRIAL: NCT01238926
Title: Effects of Vitamin Supplementation and Strength Training in Parkinson's Disease
Brief Title: Vitamin B6, B12, Folic Acid and Exercise in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Institute of Technology (Other)
Collaborators: Stony Brook University (Other)
Responsible Party: William Werner, PT, EdD, New York Institute of Technology, New York College of Osteopathic Medicine, Academic Health Care Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BHS-545
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Parkinson's Disease
Keywords: Oxidative stress; Parkinson's disease; Homocysteine; Glutathione; B vitamins
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PD vitamin supplementation (Experimental)
  Interventions: Dietary Supplement: PD vitamin supplementation
- PD exercise intervention (Experimental)
  Interventions: Other: PD exercise intervention
- PD vitamin + exercise (Experimental)
  Interventions: Other: PD vitamin + exercise
- PD control (No Intervention)

INTERVENTIONS:
Dietary Supplement: PD vitamin supplementation — 25 mg/day of Vitamin B6 2,000 mcg/day of Vitamin B12 5 mg/day of Folic Acid
  Other Names: Source Naturals® Vitamin B6 25 mg; Source Naturals® Vitamin B12 2000 mcg; Source Naturals® Folic Acid 1000 mcg
  Arms: PD vitamin supplementation
Other: PD exercise intervention — Cardiovascular training (treadmill and StairMaster), 20 min; and strength training (2 sets of 15 repetitions of 60-70% of 1 repetition maximum [RM]) using machines that provide the following motions: knee extension, knee flexion, leg press, elbow flexion, elbow extension, seated dip.
  Other Names: CYBEX(R)
  Arms: PD exercise intervention
Other: PD vitamin + exercise — 25 mg/day of Vitamin B6 2,000 mcg/day of Vitamin B12 5 mg/day of Folic Acid Cardiovascular training (treadmill and StairMaster), 20 min; and strength training (2 sets of 15 repetitions of 60-70% of 1 repetition maximum [RM]) using machines that provide the following motions: knee extension, knee flexion, leg press, elbow flexion, elbow extension, seated dip.
  Other Names: Source Naturals® Vitamin B6 25 mg; Source Naturals® Vitamin B12 2000 mcg; Source Naturals® Folic Acid 1000 mcg; CYBEX(R)
  Arms: PD vitamin + exercise

SUMMARY:
This experiment seeks to determine whether individuals with PD will benefit from vitamin B6 (pyridoxine hydrochloride), B12 (cyanocobalamin), and Folic Acid supplementation, whether they will benefit from a 6-week circuit training program, or whether they will benefit from a combination of the two interventions. The outcome variables will include: plasma homocysteine, GSH:GSSG ratio, cognitive function, balance, strength, functional activities, kinematic gait analysis, and a quality of life questionnaire.

DETAILED DESCRIPTION:
Individuals with Parkinson's disease (PD) have a higher risk of death from coronary artery disease and stroke (Gorell, Johnson, & Rybicki, 1994; Postuma & Lang, 2004). Seventy percent of people with PD suffer from dementia or cognitive impairment. Decreased levels of B vitamins are linked to increased levels of homocysteine (a protein produced in the body) which have been directly linked to heart disease, cerebrovascular accident, dementia, and impaired cognitive function (Miller et al., 2003; Postuma & Lang, 2004). Normalizing the levels of homocysteine and B vitamins in the body has been shown to reduce the risk of these diseases and improve cognitive performance (Miller et al., 2003; Morris, 2003).

Levodopa therapy, which is used to treat individuals with PD, causes elevated homocysteine levels (Blandini et al., 2001; Miller et al., 2003; Postuma & Lang, 2004). The mechanism behind the elevated homocysteine is related to vitamin B status (Miller et al., 2003; Postuma & Lang, 2004). L-dopa undergoes O-methylation and that reaction produces s-adenosylhomocysteine (SAH). SAH is then hydrolyzed and forms homocysteine. Therefore, the more L-dopa that requires 0-methylation, the more homocysteine is produced. Once homocysteine is produced, it gets metabolized back to methionine or to cysteine. In order for it to be metabolized to methionine and cysteine, Vitamin B6, B12 and Folate are needed. If homocysteine can not be metabolized, it accumulates in the body, creating dangerous levels (Miller et al., 2003; Postuma & Lang, 2004).

Undergoing levodopa therapy does not impair homocysteine metabolism but rather causes an increase in homocysteine synthesis, so that it exceeds the body's ability to metabolize it. Thus, levels of Vitamin B12 and Folate need to be higher in individuals on levodopa therapy in order to contend with the need for greater homocysteine metabolism (Miller et al., 2003).

There is ample experimental support for B vitamin supplementation to reduce homocysteine levels in this population (Lamberti et al., 2005; Miller et al., 2003; Postuma & Lang, 2004; Zoccolella et al., 2005). Supplementing B12 (cyanocobalamin) and Folic Acid have been shown to significantly decrease homocysteine levels in individuals with hyperhomocysteinemia on L-dopa therapy (Lamberti et al., 2005). Miller has shown that individuals receiving L-dopa therapy have significantly reduced levels of B6 yet normal cysteine levels. Vitamin B6 is a coenzyme in glutathione synthesis from cysteine. However, vitamin B6 (pyridoxine hydrochloride) supplementation has not been observed in this population therefore the investigators will supplement B6 as well as B12 and Folic Acid. In addition to B vitamins, exercise and strength training have been shown to lower homocysteine levels (Vincent, Bourguignon, & Vincent, 2006) and to increase resting GSH (Elokda & Nielsen, 2007).

Elevated homocysteine has been correlated with decreased glutathione levels (Mosharov, Cranford, & Banerjee, 2000). Glutathione (GSH), in part, is formed by cysteine, causing a direct link between glutathione and homocysteine (see diagram). GSH is one of the most powerful antioxidants in our body. GSH is a reduced form of glutathione which acts as our main defense against Reactive Oxygen Species (ROS) or Free Radicals (FR). ROS contribute to the initiation of many diseases (Viguie et al., 1993). Glutathione disulfide (GSSG) is the oxidized form of GSH. Typically, GSH and GSSG are measured as a ratio (GSH:GSSG) in our blood to help give an immediate understanding of the antioxidant status in our body (Elokda & Nielsen, 2007; Viguie et al., 1993). Individuals with PD have lower levels of GSH at rest than non-PD and lower levels of GSH have been directly correlated with the severity of the disease (Bharath & Andersen, 2005; Maher, 2005).

The current experiment seeks to determine if individuals with PD will benefit from supplementation of vitamins B6 (pyridoxine hydrochloride), B12 (cyanocobalamin), and folic acid, if they will benefit from a 6-week circuit training program, or if they will benefit from a combination of the two interventions. The outcome variables will include: plasma homocysteine, GSH:GSSG ratio, cognitive function, balance, strength, functional activities, kinematic gait analysis, and a quality of life questionnaire.

The investigators hypothesize that the typically lower GSH levels and higher homocysteine levels in people with PD will be normalized by supplementing B6, B12, and folate, thus reducing oxidative stress and offering more protection of ROS. The investigators hypothesize that circuit training will reduce homocysteine levels and increase glutathione levels. Furthermore, the investigators expect both interventions to improve functional measures such as gait and balance as well as improve scales measuring quality of life and depression.

Twenty-four sedentary volunteers diagnosed with PD were recruited for this study (power analysis at .80 level). All subjects were between 50 and 80 years old and rated on a Hoehn and Yahr scale at a level 2. Subjects were age and gender matched.

Each subject will perform a treadmill exercise tolerance test, and will be taken to peak exercise. Peak exercise is defined as 90% of target heart rate, an RPE of 9, if the subject is unable to maintain the pace of the treadmill, or if anaerobic threshold is attained. Additionally, the American College of Sports Medicine (ACSM) guidelines for terminating exercise testing will be followed. During the exercise test, heart rate (HR), VO2, RER, VCO2 and EKG tracings will be recorded at 1-minute intervals; BP and RPE will be recorded within the second and third minute of each stage. Vital signs, RPE and MET levels will also be recorded at termination of exercise. 3 cc of blood will be drawn immediately post exercise (within 3 minutes). The blood will be frozen and stored in a lab.

Functional Measures

Lower body functional testing will be measured by a stand-up and go timed test (Chair Stand Test) (Rikli,1999). Participants will be asked to stand from a chair and then return to sitting position. They will be asked to perform this as many times as they can in a 30 second period. It will be demonstrated by the tester first and they will be given one practice stand. There will be one 30 s trial and the total number of complete sit to stands will be the score.

Gait will be measured with kinematic analysis using a seven-camera (60 Hz) Peak Performance Motus 2000 Real-Time System (Peak Performance Technologies, Inc., Englewood, Colorado). Using a modified Helen Hayes Marker Set, passive reflective markers will be placed throughout the body allowing for precise measurement of gait (Kadaba, Ramakrishnan, & Wootten, 1990). Subjects will be asked to walk 10m along a straight, smooth, and painted concrete path. The tester will demonstrate once, and the subject will perform three trials with a seated rest of 3 min between each trial.

Balance will be tested using a SMART Balance Master System (NeuroCom International, Inc., Clackamas, Oregon). Protocols used include the Sensory Organization Test, Motor Control Test, Limits of Stability Test and the Unilateral Stance Test (Bronte-Stewart, Minn, Rodrigues, Buckley, & Nashner, 2002).

Muscle strength will be tested by joint on each individual CYBEX machine. Leg Extension, Leg Press, Leg Curl, Hip Adduction/Abduction, Rear Row, Chest Fly, Arm Curl, and Seated Dip. A one repetition maximum will be used for only one trial on each modality. The tester will perform the exercise first to demonstrate. The subject will be asked to lift as much weight as possible only one time. A 3-minute rest period will be given in between each machine.

Quality of life will be measured using the Parkinson's Disease Questionnaire 39 (PDQ-39) (Marinus, 2008 ). Psychosocial and cognitive function will be measured using the SCOPA-PS questionnaire (Marinus, Visser, Martinez-Martin, van Hilten, & Stiggelbout, 2003). Each subject will complete these questionnaires prior to the study and after completing the study.

Intervention

Blood samples, urine samples and 1 RM (ACSM Guidelines) will be measured before the exercise stress test, on the same day in the morning and fasting. Subjects will come in a second day to perform Gait analysis, balance testing, functional testing and to fill out the PDQ-39 and SCOPA questionnaire.

Each participant will be randomly assigned to one of four groups. Aerobic exercise training with weight training (AWT), AWT with B vitamin supplementation (AWT+B), B vitamin supplementation with no training (BS), and a control group (C). The exercise training sessions are 40 minutes in duration and three times per week. They will consist of 20 minutes of aerobic training either using a treadmill or an elliptical cross trainer. Since HR is not an accurate tool to determine exercise intensity in subjects with PD, participants will be monitored to maintain a HR that is consistent with V02 of 60-70% of their max V02 as determined from their initial GXT. Weight training will consist of seven CYBEX resistance exercise machines. These include leg extension, leg curl, leg press, hip abduction, latissimus dorsi pulldown, chest fly, and seated dip. Each participant will perform a 1 repetition maximum on each piece of equipment and recorded as a measure for their pre-training strength. The investigators will use 50%-80% of their 1 RM to perform 1 set of 8-15 repetitions per exercise with 30s rest period between each set of exercises (Elokda & Nielsen, 2007; Vincent et al., 2006)(ACSM). The group that is going to be supplemented will be given 5 mg/day of Folate, 2000 mcg/day of cyanocobalamin (oral B12)(Butler et al., 2006; Lamberti et al., 2005) and 25 mg/day of B6 (Malouf & Grimley Evans, 2003).

ELIGIBILITY:
Inclusion Criteria:

* Medical clearance to perform an exercise tolerance test and training program.
* A diagnosis of PD at stage 2 on the Hoehn and Yahr scale.

Exclusion Criteria:

* A neurological condition other than PD/
* Anyone who is currently taking any vitamin supplementation.
* Smokers.
* Anyone currently engaged in weight training.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Plasma homocysteine | 6 weeks
Plasma glutathione (GSH) | 6 weeks
Plasma glutathione disulfide (GSSG) | 6 weeks
GSH:GSSG ratio | 6 weeks
Plasma vitamin B6 | 6 weeks
Plasma vitamin B12 | 6 weeks
Plasma folate | 6 weeks
Balance | 6 weeks
Strength | 6 weeks
Kinematic gait analysis | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William G Werner, PT, EdD, Principal Investigator — New York Institute of Technology, New York College of Osteopathic Medicine; Joanne Donoghue, PhD, Principal Investigator — New York Institute of Technology, New York College of Osteopathic Medicine
Locations (1):
- New York Institute of Technology, New York College of Osteopathic Medicine, Academic Health Care Center, Adele Smithers Parkinson's Disease Treatment Center, Old Westbury, New York, United States

REFERENCES:
- [Background] Bronte-Stewart HM, Minn AY, Rodrigues K, Buckley EL, Nashner LM. Postural instability in idiopathic Parkinson's disease: the role of medication and unilateral pallidotomy. Brain. 2002 Sep;125(Pt 9):2100-14. doi: 10.1093/brain/awf207. PMID 12183355
- [Background] Elokda AS, Nielsen DH. Effects of exercise training on the glutathione antioxidant system. Eur J Cardiovasc Prev Rehabil. 2007 Oct;14(5):630-7. doi: 10.1097/HJR.0b013e32828622d7. PMID 17925621
- [Background] Malouf R, Grimley Evans J. The effect of vitamin B6 on cognition. Cochrane Database Syst Rev. 2003;(4):CD004393. doi: 10.1002/14651858.CD004393. PMID 14584010
- [Background] Miller JW, Selhub J, Nadeau MR, Thomas CA, Feldman RG, Wolf PA. Effect of L-dopa on plasma homocysteine in PD patients: relationship to B-vitamin status. Neurology. 2003 Apr 8;60(7):1125-9. doi: 10.1212/01.wnl.0000055899.24594.8e. PMID 12682318
- [Background] Morris MS. Homocysteine and Alzheimer's disease. Lancet Neurol. 2003 Jul;2(7):425-8. doi: 10.1016/s1474-4422(03)00438-1. PMID 12849121
- [Background] Mosharov E, Cranford MR, Banerjee R. The quantitatively important relationship between homocysteine metabolism and glutathione synthesis by the transsulfuration pathway and its regulation by redox changes. Biochemistry. 2000 Oct 24;39(42):13005-11. doi: 10.1021/bi001088w. PMID 11041866
- [Background] Postuma RB, Lang AE. Homocysteine and levodopa: should Parkinson disease patients receive preventative therapy? Neurology. 2004 Sep 14;63(5):886-91. doi: 10.1212/01.wnl.0000137886.74175.5a. PMID 15365141
- [Background] Viguie CA, Frei B, Shigenaga MK, Ames BN, Packer L, Brooks GA. Antioxidant status and indexes of oxidative stress during consecutive days of exercise. J Appl Physiol (1985). 1993 Aug;75(2):566-72. doi: 10.1152/jappl.1993.75.2.566. PMID 7693646
- [Background] Vincent HK, Bourguignon C, Vincent KR. Resistance training lowers exercise-induced oxidative stress and homocysteine levels in overweight and obese older adults. Obesity (Silver Spring). 2006 Nov;14(11):1921-30. doi: 10.1038/oby.2006.224. PMID 17135607
- [Background] Zoccolella S, Lamberti P, Armenise E, de Mari M, Lamberti SV, Mastronardi R, Fraddosio A, Iliceto G, Livrea P. Plasma homocysteine levels in Parkinson's disease: role of antiparkinsonian medications. Parkinsonism Relat Disord. 2005 Mar;11(2):131-3. doi: 10.1016/j.parkreldis.2004.07.008. Epub 2004 Dec 20. PMID 15734674